CLINICAL TRIAL: NCT04736693
Title: Replication of the HORIZON Pivotal Fracture Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-HORIZON-PFT
Record Dates: First submitted 2021-01-25; First posted 2021-02-03 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Raloxifene Hydrochloride; Zoledronic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Raloxifene: Reference Group
  Interventions: Drug: Raloxifene
- Zoledronic Acid: Exposure Group
  Interventions: Drug: Zoledronic Acid

INTERVENTIONS:
Drug: Raloxifene — Raloxifene dispensing claim is used as the reference group.
  Groups: Raloxifene
Drug: Zoledronic Acid — Zoledronic Acid dispensing claim is used as the exposure group.
  Groups: Zoledronic Acid

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Criteria:

Please see https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

Eligible cohort entry dates:

Zoledronic acid indication for treatment of postmenopausal women with osteoporosis was approved by FDA on Aug 20, 2007.

* For IBM MarketScan: Aug 21, 2007 - December 31, 2018 (end of available data)
* For Optum CDM: Aug 21, 2007 - Mar 31, 2020 (end of available data)

Inclusion Criteria:

* Postmenopausal women between the ages of 65 and 89 years
* Osteoporosis diagnosis

Exclusion Criteria:

* Bisphosphonate users
* Previous use of:

  1. Any use of parathyroid hormone
  2. Use of anabolic steroids or growth hormone within 6 months before cohort entry date OR
  3. Use of oral or intravenous systemic corticosteroids within 12 months of cohort entry date
* Serious disease that may limit life expectancy to less than 6 months
* Malignant neoplasm diagnosis within 12 months prior to the cohort entry date
* Conditions that influence bone metabolism
* Treatment and Prevention of Glucocorticoid-Induced Osteoporosis
* Treatment of Paget's Disease of Bone
* Alcohol abuse/dependence OR Drug abuse/dependence OR Non-compliance
* Pregnancy
* Diagnosis and procedure for amputee of lower limb
* Use of Zoledronic acid within 450 days prior to the cohort entry date
* Use of Denosumab within 450 days prior to the cohort entry date
* Diagnosis of End-Stage Renal Disease OR Diagnosis and procedure for Kidney transplant
* Diagnosis of End-Stage Liver Disease: Cirrhosis, Hepatic decompensation
* Blindness or compromised vision
* Use of Abaloparatide within 450 days prior to the cohort entry date
* Use of Romosozumab within 450 days prior to the cohort entry date

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Postmenopausal women with osteoporosis
Study Population: This study will involve a new user, parallel group, propensity score-matched, retrospective cohort study design comparing 15-minute annual infusions of zoledronic acid (5mg) to raloxifene. The patients will be required to have continuous enrollment during a baseline period of 450 days (15 months) before initiation of zoledronic acid or comparator. We will restrict the analyses to women, older than 65, with osteoporosis.
Sampling Method: Non-Probability Sample
Enrollment: 18028 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Number of patients with hip fracture | Through study completion (earliest of 540 days or censoring)
  Please refer to attached protocol for full definition due to size limitations

SECONDARY OUTCOMES:
Number of patients with non-vertebral fracture | Through study completion (earliest of 540 days or censoring)
  Please refer to attached protocol for full definition due to size limitations

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham And Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] D'Andrea E, Schneeweiss S, Franklin JM, Kim SC, Glynn RJ, Lee SB, Wang SV. Efficacy Versus Effectiveness: The HORIZON-Pivotal Fracture Trial and Its Emulation in Claims Data. Arthritis Rheumatol. 2025 Jan;77(1):12-21. doi: 10.1002/art.42968. Epub 2024 Sep 18. PMID 39129266

DOCUMENTS (1):
  • Study Protocol (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT04736693/Prot_001.pdf